CLINICAL TRIAL: NCT04132102
Title: An Open-label, Single-arm Clinical Study to Evaluate the Efficacy of Afatinib in Advanced Lung Squamous Cell Carcinoma With EGFR Sensitive Mutation
Brief Title: To Evaluate the Efficacy of Afatinib in Advanced Lung Squamous Cell Carcinoma With EGFR Sensitive Mutation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XK-LS-001
Record Dates: First submitted 2018-11-27; First posted 2019-10-18 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Lung Squamous Cell Carcinoma
Keywords: LSQC; EGFR mutation
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib treatment group (Experimental): This is an open-label, sing-arm phase IV clinical study
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib is a member of the second generation TKIs, which binds irreversibly to the erbB family of receptors. Afatinib will be administrated orally with the starting dose of 40 mg tablets, once per day. If patients can't tolerate drug related AEs with 40mg, patients can receive 30mg once per day after AEs recovered to Grade 0-1.
  Other Names: GIOTRIF®

SUMMARY:
This is an open-label, sing-arm, single site, phase IV clinical study. The main objective is to evaluate the efficacy of afatinib in LSQC patients with EGFR sensitive mutation, and to explore the clinical factors which might be predictive for the effectiveness in LSQC.

DETAILED DESCRIPTION:
This is an open-label, sing-arm phase IV clinical study which will recruit about 20 patients in China.

The main objective of this study is to evaluate the efficacy of afatinib in LSQC patients with EGFR sensitive mutation, and to explore the clinical factors which might be predictive for the effectiveness in LSQC.

Target patient population:Locally advanced (IIIB) or metastatic (stage IV) immunohistochemistry (IHC)-verified Lung squamous cell carcinoma (LSQC) with EGFR sensitive mutation patients, whom previously untreated or received platinum-based doublet chemotherapy as first-line treatment with subsequent disease progression, and had to be eligible for second-line treatment.

Investigational product, the dose and administration method: Afatinib is a member of the second generation TKIs, which binds irreversibly to the erbB family of receptors. Afatinib will be administrated orally with the starting dose of 40 mg tablets, once per day. If patients can't tolerate drug related AEs with 40mg, patients can receive 30mg once per day after AEs recovered to Grade 0-1 (CTCAE 5.0).

Study assessment: The collected data include the patient's demographic characteristics, information needed to determine whether the patient is eligible (including medical history, attributes of previous and current disease, and EGFR mutation status in tumor tissues), efficacy of objective response rate(ORR), progression-free survival (PFS), overall survival (OS), and safety (including serious adverse events and dose change-induced adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Selected patients must meet all of the following standards:

  1. The patient's or his/her legal representative's has signed and dated written informed consent before any specific study procedure.
  2. The patient is above 18 years old.
  3. Locally advanced (IIIB) or metastatic (stage IV) immunohistochemistry (IHC)-verified Lung squamous cell carcinoma (LSQC) with EGFR sensitive mutation patients, whom previously untreated or received platinum-based doublet chemotherapy as first-line treatment with subsequent disease progression, and had to be eligible for second-line treatment.
  4. The patient has NOT previously received EGFR-TKI treatment.
  5. ECOG Performance Status Score is 0~2.
  6. The patient has sufficient bone marrow and organ function proved by baseline complete plasma count, plasma biochemistry and urinary biochemistry tests.
  7. Female patients of childbearing age must use adequate contraceptives, and breastfeeding is not allowed.
  8. Male patients must voluntarily to use contraceptives.

     Exclusion criteria
* Selected patients can not meet any one of the following standards:

  1. The patient has received EGFR-TKI treatment.
  2. The patient has any severe or uncontrolled systemic signs of illness, including uncontrolled hypertension, active easy-bleeding constitution, active infection, or significantly impaired function of bone marrow or organs, which researchers believe can significantly change the patient's risk/benefit balance.
  3. The patient has symptomatic central nervous system (CNS) metastases.
  4. The patient has the history of interstitial pneumonia, or radiation pneumonia which needs steroid treatment.
  5. The patient still has unrecovered toxic reaction with ≥ grade 3 (CTCAE5.0) caused by previously received treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 12 months
  PFS refers to the time from initial prescription of afatinib to the time of disease progression or death recorded in CRF in this study, no matter whether the patient withdraw from the treatment before disease progression or receive other anti-cancer treatment or not. For the patient without progression or death at the time of analysis, the latest assessment date will be used as interpolation (censoring). (Or, if there's no tumor assessment after baseline visit, baseline visit date will be used

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  ORR refers to the incidence of complete remission (CR) or partial remission (PR) (determined according to RECIST1.1 standards)
Overall survival (OS) | Up to 12 months
  OS refers to the time from the patient entering into the group to the time of death. When it comes to the analysis of patients with unknown survival status, the last date when learning of the patient's survival will be used as interpolation (censoring)
Rate of SAEs, dose change-induced AEs, and AEs of particular concerns. | Up to 12 months
  Serious adverse events [SAEs], dose change-induced AEs, and AEs of particular concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Yongfeng Yu, Master, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China